CLINICAL TRIAL: NCT03094754
Title: Effect of Excised Surface Area/Body Surface Area Ratio and Location of Excision on the Postoperative Pain After Nevi Excision in Children: Observational Study
Brief Title: Excision Size and Location on the Postoperative Pain After Nevi Excision in Children
Status: Completed | Type: Observational
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Ji Eun Kim, Assitant professor, Ajou University School of Medicine
Other Study IDs: AJIRB-MED-OBS-16-533
Record Dates: First submitted 2017-03-15; First posted 2017-03-29 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Anesthesia, Endotracheal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: nevi excision — After general anesthesia, nevi excision in children is performed.

SUMMARY:
The primary purpose of this study is to investigate the effects of excised surface area/body surface area ratio and location of excision on the postoperative pain after nevi excision in children.

The primary purpose of this study is to investigate the effects of excised surface area/body surface area ratio and location of excision on the emergence excitation after nevi excision in children.

ELIGIBILITY:
Inclusion Criteria:

* children undergoing nevi excision on general anesthesia

Exclusion Criteria:

* development disorder
* neurological disorder
* psychological disorder

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: children undergoing nevi excision on general anesthesia
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2018-01-25 (Actual); Study Completion 2018-01-25 (Actual)

PRIMARY OUTCOMES:
postoperative pain score | up to 3 hours
  postoperative pain score after nevi excision

SECONDARY OUTCOMES:
emergence agitation score | up to 3 hours
  emergence agitation score after nevi excision

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Ajou University School of Medicine, Suwon, Seoum, South Korea